CLINICAL TRIAL: NCT01649791
Title: A Pilot Study of Lenalidomide as a Chemopreventive Agent for Patients With High-Risk, Early Stage B-Chronic Lymphocytic Leukemia (CLL)
Brief Title: Lenalidomide as Chemoprevention in Treating Patients With High-Risk, Early-Stage B-Cell Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 136908; NCI-2009-01327 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT01003821 (obsolete NCT alias)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Sentinel Lymph Node Biopsy; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (lenalidomide as chemoprevention) (Experimental): Patients receive lenalidomide PO once daily for 4 weeks. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Other: laboratory biomarker analysis; Procedure: lymph node biopsy; Procedure: bone marrow aspiration; Other: pharmacological study; Other: flow cytometry

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Other: laboratory biomarker analysis — Correlative study
Procedure: lymph node biopsy — Correlative study
  Other Names: Biopsy of Lymph Node
Procedure: bone marrow aspiration — Correlative study
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies
Other: flow cytometry — Correlative study

SUMMARY:
This clinical trial studies lenalidomide as chemoprevention in treating patients with high-risk, early stage B-cell chronic lymphocytic leukemia (B-CLL). Chemoprevention is the use of certain drugs to keep cancer from forming. The use of lenalidomide may slow disease progression in patients with early stage B-cell chronic lymphocytic leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine time to progression in patients with high risk CLL.

SECONDARY OBJECTIVES:

I. Overall response rate including (complete remission [CR]+partial remission [PR]) of lenalidomide.

II. To determine the incidence of immune mediated flare reaction. III. To characterize the toxicity profile of single agent lenalidomide in previously untreated B-CLL.

IV. To correlate expression of B-CLL co-stimulatory ligands and clinical efficacy of lenalidomide in this patient population.

V. To conduct correlative studies.

OUTLINE: Patients receive lenalidomide orally (PO) once daily for 4 weeks. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a definitive diagnosis of B-CLL as defined by the International Workshop on CLL (IWCll) criteria Patient must have early stage B-CLL defined as Rai stage 0, 1 or 2 Patients must not have received any prior treatment for management of B-CLL

Patients must be assessed to have high risk B-CLL as defined by either one of the following criterion:

* High-risk cytogenetics (either 17p deletion or 11q deletion);
* Unmutated immunoglobulin heavy chain gene rearrangement Patents must understand and voluntarily sign an informed consent form Able to adhere to the study visit schedule and other protocol requirements Patients must have measurable disease either an absolute lymphocyte counts (ALC) of more than 5,000/ul or measurable lymphadenopathy or organomegaly Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10-14 days prior to and again within 24 hours before starting lenalidomide and must either commit to continue abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure Able to take aspirin (81 or 325mg) or warfarin sodium daily as prophylactic anticoagulation Absolute neutrophil count >= 1.0 x 10^9/L Platelet count >= 30 x 10^9/L Serum creatinine =< 1.5 x upper limit of normal (ULN) Total bilirubin =< 1.5 mg/dL Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) < 2 x ULN or =< 5 x ULN if hepatic metastases are present

Exclusion Criteria:

Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form Pregnant or lactating females (lactating females must agree not to breast feed while taking lenalidomide) Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study Use of any other experimental drug or therapy within 28 days of baseline Known hypersensitivity to thalidomide or lenalidomide Prior history of development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs Patients who have been treated with any prior therapy for B-CLL Patients with history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off therapy for that disease for > 3 years) Patient with history of cardiac arrest within the past 6 months Any prior use of lenalidomide Concurrent use of other anti-cancer agents or treatments Known history of hepatitis B or C Known human immunodeficiency virus (HIV) positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Czuczman, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Started | 8
Completed | 5
Not Completed | 3
Not completed — Disease Progression | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients.
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Time Frame: 24 months
Population: All treated and eligible patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Number analyzed (Participants) | 8
months | 43.7 [7.6 to 43.7]

2. Secondary Outcome: Overall Response Rate (CR+PR)
Time Frame: 24 months
Population: All treated and eligible patients.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Number analyzed (Participants) | 8
percentage of participants | 100

3. Secondary Outcome: Incidence of Immune Mediated Flare Reaction
Description: Number of participants with Tumour flare.
Time Frame: 24 months
Population: All treated and eligible patients.
Measure: Number; unit: participants
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Number analyzed (Participants) | 8
participants | 4

4. Secondary Outcome: Expression of B-CLL Co-stimulatory Ligands, Mic-A, and Mic-B Assessed by Flow Cytometry
Description: PI left the institute and the data was not collected.
Time Frame: 8 days
Population: No participants were analyzed.
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Lenalidomide as Chemoprevention)
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide as Chemoprevention) (N=8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide as Chemoprevention) (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (8)
Injection site pain (General disorders) | 1 (1)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (4)
Hypersensitivity (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (3)
Ear infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood phosphorus increased (Investigations) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (8)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (3)
Hypogeusia (Nervous system disorders) | 3 (4)
Lethargy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (11)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial did not reach full accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes